CLINICAL TRIAL: NCT05481775
Title: Evaluating Anlotinib Combined With Concurrent Chemoradiotherapy Followed by Consolidation Immunotherapy Versus Concurrent Chemoradiotherapy Followed by Consolidation Immunotherapy for Locally Advanced Non-small Cell Lung Cancer: A Prospective, Randomized Controlled Phase II Clinical Trial
Brief Title: Evaluating Efficacy and Safety of Anlotinib Combined With Concurrent Chemoradiotherapy Followed by Consolidation Immunotherapy for Locally Advanced Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clincal decision based on previous results
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1088
Record Dates: First submitted 2022-07-04; First posted 2022-08-01 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Locally Advanced Non-small Cell Lung Cancer; Efficacy and Safety
Keywords: Locally advanced non-small cell lung cancer; Anlotinib combined with chemoradiotherapy; Consolidation immunotherapy
MeSH Terms: interventions — anlotinib; Drug Therapy; Chemoradiotherapy; Radiotherapy; Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): Anlotinib Combined With Concurrent Chemoradiotherapy Followed by Consolidation Immunotherapy
  Interventions: Drug: Anlotinib; Drug: Chemotherapy; Radiation: Radiotherapy; Drug: Immunotherapy
- Control group (Active Comparator): Concurrent Chemoradiotherapy Followed by Consolidation Immunotherapy
  Interventions: Drug: Chemotherapy; Radiation: Radiotherapy; Drug: Immunotherapy

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 8mg qd po. Taking anlotinib daily for 2 weeks and stop for 1 week.
  Arms: Experiment group
Drug: Chemotherapy — Docetaxel 25mg/m2 + Cisplatin 25mg/m2 QW
  Other Names: Concurrent chemoradiotherapy
Radiation: Radiotherapy — Thoracic radiotherapy was delivered using the daily image-guided intensity modulated radiation therapy (IMRT) technique. The total radiation dose was 66-68 Gy to the gross tumor in 17-22 daily fractions.
  Other Names: Concurrent chemoradiotherapy
Drug: Immunotherapy — consolidation Immunotherapy (Tislelizhu 200mg iv. drip, Q3W, up to 12 months.)

SUMMARY:
This is a prospective, randomized, controlled phase II clinical study for evaluating anlotinib combined with concurrent chemoradiotherapy followed by consolidation immunotherapy versus concurrent chemoradiotherapy followed by consolidation immunotherapy in locally advanced, unresectable NSCLC.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled phase II clinical study for evaluating anlotinib combined with concurrent chemoradiotherapy followed by consolidation immunotherapy versus concurrent chemoradiotherapy followed by consolidation immunotherapy in locally advanced, unresectable NSCLC. In this study, the enrolled patients were divided into the experimental group and the control group at a ratio of 1:1. The patients in the experimental group received anlotinib combined with curative concurrent chemoradiotherapy first, while the patients in the control group received curative concurrent chemoradiotherapy. Those who are evaluated as CR, PR or SD after the aforementioned treatment will enter consolidation immunotherapy. Patients will receive tislelizumab 200mg iv. drip, Q3W, for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* informed consent is required before proceeding with any steps in the study;
* Male or female 18-75 years old;
* Patients must be locally advanced, unresectable (stage IIIA-IIIC) with histology reported NSCLC (except for central squamous cell carcinoma or those at risk for massive hemoptysis);
* No prior chemotherapy, immunotherapy, radiotherapy, surgery, or targeted therapy;
* Tumor sample requirements: must provide sufficient evidence to allow analysis Stained, archived tumor tissue samples;
* Life expectancy ≥ 12 weeks;
* World Health Organization (WHO) PS score of 0 or 1;
* Postmenopausal women, or negative urine or serum pregnancy test (HCG) within 14 days prior to study drug administration
* Women of childbearing potential (WOCBP) must agree to adhere to contraceptive methods during study drug treatment and for 6 months after the last study drug treatment;
* Men who have sex with WOCBP must agree to adhere to contraception during study drug treatment and for 6 months after the last study drug treatment;
* azoospermic men do not have to adhere to contraceptive requirements. Adolescents of childbearing potential without heterosexual sex (WOCBP) do not have to comply with contraceptive requirements, but must still undergo a pregnancy test as described in this section;
* Organ and bone marrow function meet the following conditions: Forced expiratory volume in 1 second (FEV1) ≥ 800ml; Absolute neutrophil count ≥1.5×10^9/L; Platelet ≥100×10^9/L; Hemoglobin ≥9.0g/dL; Serum creatinine clearance calculated according to Cockcroft-Gault formula ≥50 mL/ min (Cockcroft and Gault 1976); Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN); AST and ALT ≤ 2.5 times ULN.

Exclusion Criteria:

* Concurrent participation in another clinical study, unless it is an observational (non-interventional) clinical study;
* Histological type of small cell lung cancer (including mixed small cell and non-small cell lung cancer);
* Prior use of any targeted therapy;
* The central cavity squamous cell carcinoma or non-small cell lung cancer with hemoptysis (the amount of hemoptysis> 50 ml/d);
* The patient has conditions that affect oral medication (such as dysphagia, chronic diarrhea, intestinal obstruction, etc.) ;
* Major surgery (excluding vascular access) within 4 weeks prior to study entry;
* Heart rate-corrected mean QT interval (QTc) ≥ 470 ms, calculated from 3 electrocardiogram calculation cycles (ECG) using Bazett correction;
* No Controlled complications, including but not limited to persistent or active infection, symptomatic congestive heart failure, poorly controlled hypertension, unstable angina, arrhythmia, active peptic ulcer disease or gastritis, active hemorrhagic Illness, including any known HBsAg-positive patient with HBV DNA > 500 IU/ml, Hepatitis C or Human Immunodeficiency Virus (HIV), or mental illness that would limit compliance with study requirements or impair the patient's ability to give written informed consent/ Social status;
* History of another primary malignancy within 5 years prior to initiation of therapy, excluding adequately treated skin basal or squamous cell carcinoma or cervical carcinoma in situ;
* Pregnant, breastfeeding women; Contraceptive method, male or female of reproductive potential; - Conditions that may interfere with the evaluation of the efficacy or safety of the treatment.
* Patients who progressed after concurrent chemoradiotherapy;
* History of tuberculosis, excluding old pulmonary tuberculosis;
* Received live attenuated vaccine within 30 days before study initiation or within 30 days after tislelizide;
* In Use of immunosuppressive drugs within 28 days prior to the first dose of tislelizumab. Of these, intranasal inhaled corticosteroids at physiological doses are excluded; prednisone or an equivalent amount of systemic corticosteroids not exceeding 10 mg per day is excluded. Steroids are permitted for management of chemoradiotherapy-related toxicity;
* Patients with unrecovered CTCAE > 2 toxicity after prior targeted combination chemoradiotherapy will be excluded from randomization;
* due to prior targeted combined chemoradiotherapy, patients with grade ≥2 pneumonitis undergoing chemotherapy will be excluded from randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
18-months progression-free survival rate | 18-months
  From the first day of treatment to the day of progression or the day of death.

SECONDARY OUTCOMES:
Overall survival | 18-months
  It was calculated from the first day of treatment to the day of death.
objective response rate | 18-months
  The proportion patients evaluated for CR and PR
Incidence of Treatment-related Adverse Events | 18 months after therapy
  Adverse effects are graded according to the CTCAE 5.0 version, including multiple organs and tissues, such as gastrointestinal disease and symptom, cardiovascular disease, respiratory diseases and so on.
Score of EORTC QLQ-C30 | 18 months after therapy
  The evaluation of life quality

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Faivre-Finn C, Vicente D, Kurata T, Planchard D, Paz-Ares L, Vansteenkiste JF, Spigel DR, Garassino MC, Reck M, Senan S, Naidoo J, Rimner A, Wu YL, Gray JE, Ozguroglu M, Lee KH, Cho BC, Kato T, de Wit M, Newton M, Wang L, Thiyagarajah P, Antonia SJ. Four-Year Survival With Durvalumab After Chemoradiotherapy in Stage III NSCLC-an Update From the PACIFIC Trial. J Thorac Oncol. 2021 May;16(5):860-867. doi: 10.1016/j.jtho.2020.12.015. Epub 2021 Jan 19. PMID 33476803
- [Result] Lin B, Song X, Yang D, Bai D, Yao Y, Lu N. Anlotinib inhibits angiogenesis via suppressing the activation of VEGFR2, PDGFRbeta and FGFR1. Gene. 2018 May 15;654:77-86. doi: 10.1016/j.gene.2018.02.026. Epub 2018 Feb 14. PMID 29454091
- [Result] Palakurthi S, Kuraguchi M, Zacharek SJ, Zudaire E, Huang W, Bonal DM, Liu J, Dhaneshwar A, DePeaux K, Gowaski MR, Bailey D, Regan SN, Ivanova E, Ferrante C, English JM, Khosla A, Beck AH, Rytlewski JA, Sanders C, Laquerre S, Bittinger MA, Kirschmeier PT, Packman K, Janne PA, Moy C, Wong KK, Verona RI, Lorenzi MV. The Combined Effect of FGFR Inhibition and PD-1 Blockade Promotes Tumor-Intrinsic Induction of Antitumor Immunity. Cancer Immunol Res. 2019 Sep;7(9):1457-1471. doi: 10.1158/2326-6066.CIR-18-0595. Epub 2019 Jul 22. PMID 31331945
- [Result] Yang Y, Li L, Jiang Z, Wang B, Pan Z. Anlotinib optimizes anti-tumor innate immunity to potentiate the therapeutic effect of PD-1 blockade in lung cancer. Cancer Immunol Immunother. 2020 Dec;69(12):2523-2532. doi: 10.1007/s00262-020-02641-5. Epub 2020 Jun 23. PMID 32577817
- [Result] Liu S, Qin T, Liu Z, Wang J, Jia Y, Feng Y, Gao Y, Li K. anlotinib alters tumor immune microenvironment by downregulating PD-L1 expression on vascular endothelial cells. Cell Death Dis. 2020 May 4;11(5):309. doi: 10.1038/s41419-020-2511-3. PMID 32366856
- [Result] Guo L, Zhang L, Guan Y, Li Y, Zhang C, Guo Q. In vitro studies of H520 cell cycle and apoptosis by anlotinib combined with radiotherapy. Thorac Cancer. 2021 Mar;12(5):593-602. doi: 10.1111/1759-7714.13780. Epub 2021 Jan 12. PMID 33438349
- [Result] He Z, Liu J, Ma Y, Jiang H, Cui Z, Wang G, Wu Y, Liu J, Cai X, Qian J, Huang J, Zhang H, Li H. Anlotinib Combined with Cranial Radiotherapy for Non-Small Cell Lung Cancer Patients with Brain Metastasis: A Retrospectively, Control Study. Cancer Manag Res. 2021 Aug 4;13:6101-6111. doi: 10.2147/CMAR.S319650. eCollection 2021. PMID 34377028
- [Result] Zhuang H, Wang Y, Cheng C, Shi S. The efficacy of anlotinib instead of glucocorticoids for edema induced by brain metastases in NSCLC patients with anti-PD1/PDL-1 immunotherapy. Neuro Oncol. 2021 Jan 30;23(1):169-171. doi: 10.1093/neuonc/noaa236. No abstract available. PMID 33294918
- [Result] Wang Y, Deng W, Li N, Neri S, Sharma A, Jiang W, Lin SH. Combining Immunotherapy and Radiotherapy for Cancer Treatment: Current Challenges and Future Directions. Front Pharmacol. 2018 Mar 5;9:185. doi: 10.3389/fphar.2018.00185. eCollection 2018. PMID 29556198
- [Result] Liao ZX, Komaki RR, Thames HD Jr, Liu HH, Tucker SL, Mohan R, Martel MK, Wei X, Yang K, Kim ES, Blumenschein G, Hong WK, Cox JD. Influence of technologic advances on outcomes in patients with unresectable, locally advanced non-small-cell lung cancer receiving concomitant chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):775-81. doi: 10.1016/j.ijrobp.2009.02.032. Epub 2009 Jun 8. PMID 19515503
- [Result] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Result] Franceschini D, Paiar F, Meattini I, Agresti B, Pasquetti EM, Greto D, Bonomo P, Marrazzo L, Casati M, Livi L, Biti G. Simultaneous integrated boost-intensity-modulated radiotherapy in head and neck cancer. Laryngoscope. 2013 Dec;123(12):E97-103. doi: 10.1002/lary.24257. Epub 2013 Jun 26. PMID 23775348
- [Result] Wu B, McNutt T, Zahurak M, Simari P, Pang D, Taylor R, Sanguineti G. Fully automated simultaneous integrated boosted-intensity modulated radiation therapy treatment planning is feasible for head-and-neck cancer: a prospective clinical study. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):e647-53. doi: 10.1016/j.ijrobp.2012.06.047. Epub 2012 Aug 3. PMID 22867890